CLINICAL TRIAL: NCT02103283
Title: Phase 1, Open-Label Safety and Pharmacodynamic Study of RV001, an Insulin-Like Growth Factor-1 Receptor (IGF-1R) Antagonist, Administered by Intravenous (IV) Infusion in Patients With Diabetic Macular Edema (DME)
Brief Title: A Phase 1, Open-Label Study of Teprotumumab in Patients With Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DME01RV
Record Dates: First submitted 2014-03-27; First posted 2014-04-03 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema
MeSH Terms: interventions — teprotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teprotumumab (Experimental): Teprotumumab 20mg/kg administered by intravenous infusion every 3 weeks for 3 infusions
  Interventions: Drug: Teprotumumab

INTERVENTIONS:
Drug: Teprotumumab — Teprotumumab 20mg/kg administered by intravenous infusion every 3 weeks for 3 infusions
  Other Names: RV 001

SUMMARY:
A Phase 1 Study to evaluate the Safety of teprotumumab in Patients with Diabetic Macular Edema.

DETAILED DESCRIPTION:
A Phase 1, Open-Label Safety and Pharmacodynamic Study of RV 001, an Insulin-Like Growth Factor-1 Receptor (IGF-1) Antagonist, Given By IV Infusion in Patients with Diabetic Macular Edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus with Hemoglobin A1c <8.5%
* IGF 1 in serum > 106 ng/mL
* Women of child-bearing potential must have negative pregnancy test and be willing and able to use two different methods of contraception, one of which must be oral contraceptive or depot formulation. Males must be surgically sterile or agree to use barrier contraception
* Clinically significant DME of less than 12 months duration
* Non-proliferative diabetic retinopathy of moderate severity
* Best corrected electronic ETDRS letter score < 78 and > 24

Exclusion Criteria:

* Unstable-uncontrolled diabetes as demonstrated by a change in diabetes medication greater than 15% in the previous 60 days.
* Significant renal disease, myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure
* Blood pressure > 180/110
* Anti-vascular endothelial growth factor (VEGF) treatment within two months prior to enrollment
* History of pan retinal photocoagulation within four months prior to enrollment
* History of ocular surgery within four months prior to enrollment
* History of systemic treatment with corticosteroids within 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety of RV001in subjects with Diabetic Macular Edema | Change from Baseline to Week 9
  Number of subjects with adverse events, serious adverse events and early discontinuations due to adverse events. Number of subjects with clinical significant abnormal laboratory values, electrocardiograms (pre and post infusions), abnormal vital signs, ophthalmic and physical examinations.

SECONDARY OUTCOMES:
Safety of RV001in subjects with Diabetic Macular Edema | Change from Baseline to Week 9
  Pharmacodynamic measure includes change in Optical Coherence Tomography, Fluorescein Angiography and Stereoscopic color funds photos findings.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - David S Boyer, Beverly Hills, California
  - David A Eichenbaum, MD, St. Petersburg, Florida
  - Diana Do, MD, Omaha, Nebraska